CLINICAL TRIAL: NCT05999175
Title: Evaluation of the Tolerability, Safety of Use, and Efficacy of Cosmetic Products for the Oral Care. In Use Test Under Dentist Control
Brief Title: Open-label Trial Evaluating Four Oral Hygiene Regimens Using a Manual Toothbrush, Toothpaste, and Mouthwash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biokosmes Srl (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0002847/21
Record Dates: First submitted 2023-07-20; First posted 2023-08-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Oral Hygiene; Toothbrushing; Dental Plaque
Keywords: Gingival sensitivity; manual toothbrush; mouthwash; oral hygiene; oral microbiota stability; oral mucosa; plaque reduction; toothbrush; toothpaste
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Study participants would be randomly allocated to one of the following groups: Group 1 (20 subjects) would use the delicate mint toothpaste "Dentifricio gel tau-marin® Menta Delicata"; Group 2 (12 subjects) mint toothpaste " Dentifricio gel tau-marin® Menta"; Group 3 (20 subjects) mint mouthwash "Collutorio tau-marin® Menta". Group 4 (20 subjects) would utilize delicate mint toothpaste "Dentifricio gel tau-marin® Menta Delicata" and mint mouthwash " Collutorio tau-marin® Menta". These products would be applied with tau-marin® scalar toothbrush 33 medium with antibacterial "Spazzolino tau-marin®" three times a day after the main meals for 28 days. Group 5 (12 subjects) would continue to use routine oral hygiene products for 28 days. Groups 1 to 3 would be provided with a standard toothbrush (without any claims of efficacy) to be used three times a day after the main meals for 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (20 subjects) (Other): using the delicate mint toothpaste "Dentifricio gel tau-marin® Menta Delicata".
  Interventions: Device: the toothpaste is used with a standard toothbrush without any claims 3 times a day after the main meals for 28 days.
- Group 2 (12 subjects) (Other): using of the mint toothpaste "Dentifricio gel tau-marin® Menta".
  Interventions: Device: the toothpaste is used with a standard toothbrush without any claims 3 times a day after the main meals for 28 days.
- Group 3 (20 subjects) (Other): using the mint mouthwash "Collutorio tau-marin® Menta.
  Interventions: Device: the toothpaste is used with a standard toothbrush without any claims 3 times a day after the main meals for 28 days.
- Group 4 (20 subjects) (Other): using the delicate mint toothpaste "Dentifricio gel tau-marin® Menta Delicata", mint mouthwash "Collutorio tau-marin® Menta".
  Interventions: Device: the mint toothpaste and mouthwash are used with the scalar toothbrush 33 medium with antibacterial " Spazzolino tau-marin®" 3 times a day after the main meals for 28 days.
- Group 5 (12 subjects) (Other): continuing to use their routine oral hygiene products.
  Interventions: Device: subjects of this group will use their routine oral hygiene products.

INTERVENTIONS:
Device: the toothpaste is used with a standard toothbrush without any claims 3 times a day after the main meals for 28 days. — the toothpaste is used with a standard toothbrush without any claims 3 times a day after the main meals for 28 days.
  Arms: Group 1 (20 subjects); Group 2 (12 subjects); Group 3 (20 subjects)
Device: the mint toothpaste and mouthwash are used with the scalar toothbrush 33 medium with antibacterial " Spazzolino tau-marin®" 3 times a day after the main meals for 28 days. — the mint toothpaste and mouthwash are used with the scalar toothbrush 33 medium with antibacterial " Spazzolino tau-marin®" 3 times a day after the main meals for 28 days.
  Arms: Group 4 (20 subjects)
Device: subjects of this group will use their routine oral hygiene products. — subjects of this group will use their routine oral hygiene products.
  Arms: Group 5 (12 subjects)

SUMMARY:
The purpose of this open-label, randomized controlled clinical trial, is to provide preliminary clinical data (efficacy on plaque and gingival sensitivity, and safety and tolerability of two types of toothpaste, a mouthwash, and a specifically custom-designed toothbrush used for 28 days), as well as descriptive data on the effects of the products on oral microbiota rebalancing and patient acceptability. Eighty-four participants with a history of poor oral hygiene are visited at baseline and after 28 days of administration of the tested products. The control group consisted of 12 participants who continued to use their oral care products without changing their normal routine. At baseline and at the end of treatment (final visit), the oral microbiome is also evaluated in a group of 12 subjects allocated randomly.

DETAILED DESCRIPTION:
A complete line of cosmetic products (Tau-marin Protezione e Prevenzione) was launched on the Italian market in 2023. These products are based on an innovative formulation containing a prebiotic (Bioecolia®) and a paraprobiotic based on Lactobacillus plantarum (SymrebootTM OC). The products are the toothpastes "Dentifricio Menta Delicata" and "Dentifricio Menta" and the mouthwash "Collutorio Menta". The products should preferably be used with the "Spazzolino tau-marin" toothbrush, which, thanks to the silver ions placed on the bristles, handle and head of the toothbrush, can eliminate Staphylococcus aureus, methicillin-resistant Staphylococcus aureus (MRSA), Pseudomonas aeruginosa and Escherichia coli bacteria. Bioecolia® is an alpha-glucan oligosaccharide that is a preferred substrate for commensal bacteria and selectively stimulates their growth. SymrebootTM OC belongs to the class of paraprobiotics, i.e. non-viable microbial cells (either intact or disrupted) or crude cell extracts, which, when administered in adequate amounts, provide a health benefit to the user. SymrebootTM OC consists of heat treated Lactobacillus plantarum HEAL19. The combined action of prebiotic and paraprobiotic results in the restoration of the symbiosis. Stability and preclinical tests confirm the safety of these products for oral hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males and females aged ≥ 18 to ≤ 65 years included.
* Proper oral hygiene not performed verified with Simplified Oral Hygiene Index (OHI-S) (score ≥ 2) and a questionnaire on oral habit.
* Patients able to comply with the requirements for the study and freely willing to provide written informed consent to the collection of their data.
* Registered with Italian National Health Service (NHS).
* Ability to understand the language used in the investigation center and to comply with the study procedures.
* Unbanned pharmacological therapy stable for at least one month without any changes during the study.
* Commitment not to change the daily routine and lifestyle.

Exclusion Criteria:

* Allergies or sensitivity to oral care products, cosmetic products, drugs, patch or medical devices.
* Any oral cavity condition inappropriate for participation.
* Gums bleeding due to pathologies/pharmacological treatment.
* Concomitant or during the last week antibiotic therapy.
* Smokers (≥5 cigarettes/day).
* Acute, chronic or progressive diseases/illness/conditions able to interfere with the outcome of the study or considered dangerous or incompatible with the study requirements.
* Pathological staining of teeth.
* Breast-feeding, pregnancy, or women of child-bearing age unwilling to take the necessary precautions to avoid pregnancy during the study.
* Planning to participate or participation in other clinical trials withing 30 days.
* Hospitalization/planned hospitalization in a health or social facility.
* Deprivation of freedom by administrative or legal decision or under guardianship
* Inability to be contacted in case of emergency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Gums sensitivity | 28 days
  Change from baseline to day 14 and 28 days assessed by the Investigator during the dentist examination using a 10 cm visual analogue scale (VAS) where 0 is absence of sensitivity and 10 indicates the maximum of sensitivity.
Rate of gingival irritations | 28 days
  Change from baseline to 14 and 28 days assessed by the Investigator during the dentist examination as follows: (Yes presence of gingival irritation; No = absence of gingival irritation).
Rate of oral mucosa lesions | 28 days
  Change from baseline to 14 and 28 days assessed by the Investigator during the dentist examination as follows: (Yes presence of oral mucosa lesion; No = absence of oral mucosa lesion).
Dental plaque assessment | 1 day
  Change from T0 (at the baseline at visit, performed three hours after the last teeth brushing) to Timm (evaluation done immediately after the first product use). The evaluation is carried out by means of an erythrosine-based disclosing tablet, which allows to quantify the presence of plaque on the teeth. First, the dentist gives the tablet to the subjects, who are asked to chew it thoroughly in their mouths. Then, the subjects are asked to rub the chewed particles of the tablets on their teeth with their tongue and swish the accumulated saliva in their mouth for about 60 seconds before rinsing with water. The releasing tablet stains the plaque on the teeth.
Teeth colour assessment | 28 days
  Change from baseline to 14 and 28 days as assessed by the investigator during the dentist's examination comparing the subjects' teeth with those shown on the VITAPAN® Score. The scoring system consists of a series of 16 "artificial teeth" in 16 different colors, each of which is associated with an alphanumeric code representing the entire chromatic space of natural teeth. It classifies tooth color into 4 families of shades as follows: reddish-brownish (A1, A2, A3, A3.5, A4), reddish-yellowish (B1, B2, B3, B4), grayish (C1, C2, C3, C4) and reddish-grey (D2, D3, D4).

SECONDARY OUTCOMES:
Self-assessment questionnaire | 28 days
  Subjects are asked to complete a self-report questionnaire on Timm (immediately after first use) and on days 14 and 28.
Oral microbiota analysis | 28 days
  It evaluates the change from baseline to 28 days. Oral microbiota is obtained by brushing a defined area of the mouth. Swabs are collected and stored at room temperature. Microbiome analysis is based on metagenomic analysis of the 16S rRNA gene.
  The second step in the analysis pipeline is to isolate the bacterial DNA from other components of the sample. Through a series of cell lysis and extraction steps, the purified bacterial material is obtained. The bacterial material is then amplified by PCR, first to increase the amount of DNA, and second to label the genetic material - which will later allow identification of each sample during the sequencing step. The concentrations of the samples are equalized prior to pooling to create the sequencing mix. This solution is then loaded into a cartridge and analyzed by a sequencer. The biodiversity index (Shannon index) and statistics are calculated using a dedicated software (Microbiome analyst)
Serious Adverse Events/Adverse Events | 14 days
  The number of participants with treatment-related adverse events will be assessed by CTCAE v6.0

CONTACTS AND LOCATIONS:
Overall Officials: Dario Cattaneo, DDS, Principal Investigator — San Genesio ed Uniti, Pavia (Italy)
Locations (2):
- Italy (2):
  - Studio D. Cattaneo, San Genesio ed Uniti, Pavia
  - Complife Italia Srl, San Martino Siccomario, Pavia

REFERENCES:
- [Background] Willis JR, Gabaldon T. The Human Oral Microbiome in Health and Disease: From Sequences to Ecosystems. Microorganisms. 2020 Feb 23;8(2):308. doi: 10.3390/microorganisms8020308. PMID 32102216
- [Background] Abdulkareem AA, Al-Taweel FB, Al-Sharqi AJB, Gul SS, Sha A, Chapple ILC. Current concepts in the pathogenesis of periodontitis: from symbiosis to dysbiosis. J Oral Microbiol. 2023 Apr 2;15(1):2197779. doi: 10.1080/20002297.2023.2197779. eCollection 2023. PMID 37025387
- [Background] Kilian M, Chapple IL, Hannig M, Marsh PD, Meuric V, Pedersen AM, Tonetti MS, Wade WG, Zaura E. The oral microbiome - an update for oral healthcare professionals. Br Dent J. 2016 Nov 18;221(10):657-666. doi: 10.1038/sj.bdj.2016.865. PMID 27857087
- [Background] Rajendiran M, Trivedi HM, Chen D, Gajendrareddy P, Chen L. Recent Development of Active Ingredients in Mouthwashes and Toothpastes for Periodontal Diseases. Molecules. 2021 Apr 1;26(7):2001. doi: 10.3390/molecules26072001. PMID 33916013
- [Result] Rosu S, Benatti P, Bianco S, Barattini DF, Nobile V, Mellai M, Cattaneo D. Pilot, open-label, randomized controlled clinical trial evaluating 4 oral hygiene regimens using a manual toothbrush, toothpaste, and mouthwash. Gen Dent. 2024 Jul-Aug;72(4):62-71. PMID 38905608
- See also: Bioecolia® is the prebiotic included in the tested products. — https://www.solabia.com/cosmetics/product/bioecolia/